CLINICAL TRIAL: NCT06790589
Title: COmparison of Two Alternative Thyrotropin Suppression Strategies Among Patients With Advanced Differentiated Cancer of the tHyroid
Brief Title: COACH - Comparing Two Different Methods to Suppress Thyrotropin in Patients With Advanced Thyroid Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0033
Record Dates: First submitted 2025-01-09; First posted 2025-01-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Differentiated Thyroid Gland Carcinoma
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levothyroxine dosing with a target Thyrotropin (TSH) suppressed level of <0.1 mU/L (Active Comparator): Levothyroxine oral tablet treatment daily with doses optimized to achieve an initial target TSH level of <0.1 mU/L for a total of two years.
  Interventions: Drug: Levothyroxine Oral Tablet [Synthroid]
- Levothyroxine dosing with a target Thyrotropin (TSH) suppressed level of 0.1 - 0.5 mU/L (Experimental): Levothyroxine oral tablet treatment daily with doses optimized to achieve an initial target TSH level of 0.1-0.5 mU/L for a total of two years.
  Interventions: Drug: Levothyroxine Oral Tablet [Synthroid]

INTERVENTIONS:
Drug: Levothyroxine Oral Tablet [Synthroid] — Round, colour coded, scored tablet debossed with "SYNTHROID" on one side and potency on the other side.

SUMMARY:
Most thyroid cancers can be cured with surgery, sometimes with radioactive iodine therapy. However, some patients have cancer that has spread, and some have cancer that comes back after treatment. For those with remaining cancer, lowering TSH levels is recommended. This is because thyroid cancer growth can depend on TSH, so reducing TSH can lower the risk of cancer returning and slow its growth in patients with cancer that can't be surgically removed.

International guidelines recommend keeping TSH levels as low as <0.1 mU/L for patients with advanced thyroid cancer. This advice is based on past studies, but it hasn't been tested in a controlled way. One old study suggested that not lowering TSH enough could lead to more cancer relapses. Another study suggested that lowering TSH more could help prevent cancer from getting worse in high-risk patients. However, a recent study found no link between TSH levels and better outcomes, and the researchers suggested doing a new study to confirm if this practice is truly beneficial.

Lowering TSH levels to <0.1 mU/L using levothyroxine has been the standard of care for treating advanced thyroid cancer for a long time. The researchers would like to investigate whether using levothyroxine to keep TSH levels between 0.1 and 0.5 mU/L is just as safe and effective for cancer treatment as the current recommendation of keeping it below 0.1 mU/L. The researchers also believe this study can help set TSH suppression targets based on cancer type, reducing unnecessary side effects from too much TSH suppression while still achieving the same cancer treatment results.

If the researchers can prove that keeping TSH levels between 0.1 and 0.5 mU/L is just as safe and effective as the standard of care practice, we can change our standard treatment approach. This would help reduce symptoms for our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age of 18 years, with no upper limit of age.
2. ECOG 0-2
3. Patients must be capable of providing consent to enrollment and willing to comply with study treatment and follow-up.
4. Diagnosis of differentiated thyroid cancer (including papillary, follicular, oncocytic, and poorly differentiated subtypes) with advanced structural disease (defined as unresectable persistent/ recurrent locoregional disease and/or distant metastases).
5. Residence within Alberta and referral to the Cross Cancer Institute in Edmonton, for consideration of anticancer therapy and/or follow-up.
6. Absence of any condition hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the study.
7. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 30 days after the last dose of study drug. A highly effective method of birth control is defined as those resulting in low failure rate (i.e., less than 1% per year) when used consistently and correctly.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient.
8. Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
9. Females must not be breastfeeding (timeframe: during study treatment period and for a period of 30 days after the last dose of the study drug).
10. Ability to obtain sufficient thyroid cancer tissue to conduct baseline NGS testing (could be fresh or archived tissue).

Exclusion Criteria:

1. Recent acute coronary event (within 6 months of randomization).
2. History of atrial fibrillation.
3. Known hypersensitivity to levothyroxine.

   - Treatment with other investigational drugs within 30 days prior to randomization.
4. History of fragility fractures or established diagnosis of osteoporosis.

   * Prior treatment with levothyroxine before study entry at any dose and with any TSH target is not an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Who are Alive and Progression-free at One Year | up to 1 year after randomisation.
  Progression will be defined using RECIST criteria 1.1 and will be based on radiological assessment only. Biomarkers (such as thyroglobulin) will not be considered given the significant limitations associated with these biomarkers in the setting of locally recurrent or metastatic differentiated thyroid cancer.

SECONDARY OUTCOMES:
Mean Change of Symptom Burden (as assessed by ESAS) | Screening, 6 months, 12 months, 18 months, 24 months
  Edmonton Symptom Assessment Score (ESAS) is a standard way of monitoring patient-reported outcomes in all Cancer Care Alberta facilities. Through this system, we will assess the trajectory of symptom burden across preplanned timepoints during the study duration. We will add hyperthyroidism-specific symptoms (e.g., racing heart or palpitations) in the others category of the ESAS form.
Proportion of Patients Who are Alive and Progression-free at One Year According to Molecular Subtype (RAS-like vs BRAF-like cancers) | 1 year after randomization
  Cancers with the following molecular changes within initial NGS, will be considered as BRAF-like (BRAF V600E mutation, NTRK fusion, ALK fusion, and RET fusion). Cancers with the following molecular changes will be considered as RAS-like (any RAS mutation, BRAF 601E, PAX 8/PPARG). We will examine if there is a difference in the oncological impact of TSH suppression among patients with BRAF-like tumors vs those with RAS-like tumors (given the clinical and biological differences between these two groups of patients). This outcome will be measured one year after randomization.
  NGS testing is currently conducted by Alberta Precision Labs and should be funded from the study's budget (for patients who have not had testing already prior to study entry as part of their routine clinical care).
Median Progression-free Survival | 6 months, 12 months or death
  Progression-free survival is defined as the time from randomization until radiological disease progression or death. Assessment of progression will be based only on RECIST criteria version 1.1.
Rate of levothyroxine-related adverse events | Screening to End of Study (2 years)
  We would like to examine the difference between levothyroxine-related adverse events in both groups (including diarrhea, anxiety, psychiatric disorders, cardiac adverse events, among others). We will report all grade adverse events comparing the number of AEs between each group.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abdelsalam, Principal Investigator — Cross Cancer Institute